CLINICAL TRIAL: NCT01054911
Title: Pilot Trial of Neoadjuvant Sunitinib in Patients With Bulky GIST
Brief Title: Evaluation of Patients With Bulky GIST Using Sunitinib
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor accrual
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, James Posey, MD, Associate Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F090910001; UAB 0855 (Other: Institutional study protocol number)
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-08

CONDITIONS: Tumor
Keywords: GIST; gastrointestinal stromal tumor; gastrointestinal stomach tumor; Sunitinib
MeSH Terms: conditions — Neoplasms; Gastrointestinal Stromal Tumors | interventions — Sunitinib; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib pill (Experimental): Patients will receive six weeks of sunitinib and then subsequently continue for an additional 6 weeks if the evaluation at 6 weeks shows stable disease or objective response. Restaging CT scans will be performed again after 12 weeks of therapy to determine response in preparation for surgical resection anticipated to occur around week 14-16.
  Interventions: Drug: Sunitinib; Procedure: Surgery

INTERVENTIONS:
Drug: Sunitinib — All patients will receive sunitinib 37.5 mg p.o. daily for up to 12 weeks to be taken orally.
  Other Names: SUTENT (Sunitinib)
Procedure: Surgery — Following sunitinib therapy, patients will be evaluated for surgery. It is anticipated that the quality of response will allow for complete resection of residual tumor. Surgical resection, if eligible, will occur around week 14-16.

SUMMARY:
The primary purpose of this study is to determine if oral (mouth) delivery prior to tumor removal in patients with gastrointestinal stromal tumor (GIST) results in tumor shrinkage allowing for successful surgery. Therapy will be administered orally and the response of the tumor will be assessed using CTs or MRIs.

DETAILED DESCRIPTION:
Gastrointestinal stromal tumor (GIST) is a rare cancer affecting primarily the digestive tract and sometimes abdominal cavity in adults. The most common site is the stomach followed by the duodenum and small intestine.

Surgery is the mainstay of therapy for GIST patients whose primary tumor is felt to be resectable. Prior to the introduction of Gleevec, patients with inoperable GIST had essentially no therapeutic options. However, sunitinib trials offer options to patients who are Gleevec resistant or have intolerant GIST. Clinical benefit has been demonstrated with positive results in several sunitinib studies of varying phases.

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 19 years old with pathologically proven GIST which is bulky or marginally resectable
* Patients must have at least one bidimensionally measurable disease site of 5 cm or greater not previously irradiated. Bone lesions do not qualify.
* Patients must have an ECOG performance of greater than or equal to 2, with projected survival of at least three months.
* Patients must have adequate laboratory parameters:

Hematologic: Hb >9.0; WBC >3200 and platelets >100,000/mm3; Hepatic: Bilirubin <2.0 and AST within 4 times upper limit of normal; Renal: Creatinine of less than or equal to 1.6 or eGFR greater than or equal to 50 mL/min

* Men and women who are of childbearing potential must practice strict birth control for the duration of the study.
* Women of childbearing potential must be non-lactating and non-pregnant with a negative pregnancy test within two weeks of trial registration.
* The patient, a witness, and attending physician will have signed an IRB-approved informed consent prior to Sunitinib administration.

Exclusion Criteria:

* Known brain metastases or significant pleural effusion or ascites.
* Uncontrolled hypertension, diabetes, or other medical condition.
* Major surgery within 21 days of registration.
* Patients wtih organ grafts with the exception of prior high dose chemotherapy with autologous bone marrow (or stem cell) transplantation.
* History of seizures, central nervous system disorders, dementia, or psychosis that might preclude adequate informed consent or protocol compliance.
* Prior therapy for GIST.
* A history of HIV or hepatitis virus infection.
* Any recent medical condition which, in the opinion of the investigator, makes the patient unsuitable for study participation.
* Patients with impaired kidney function.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A. Posey, M.D., Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sunitinib Pill
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Gastrointestinal stromal tumor comprise 1% of gastrointestinal tumors. There are 6000 new cases per year in the United States without apparent geographic, ethnic, or gender prevalence.
Arm/Group | Sunitinib Pill
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: 6 months
Measure: Number; unit: participants
Groups:
- Neoadjuvant Therapy Plus Surgery: Patients received oral therapy for up to 12 weeks and re-evaluated for response. Favorable tumor reduction resulted surgical extirpation typically with less morbid operative intervention.
- Neoadjuvant Therapy no Surgery: Patients received oral therapy for up to 12 weeks. Reassessment demonstrated response, but no surgical intervention
Arm/Group | Neoadjuvant Therapy Plus Surgery | Neoadjuvant Therapy no Surgery
Number analyzed (Participants) | 4 | 1
participants | 4 | 1

2. Secondary Outcome: Measurable Disease Response Rate
Description: Positron electron emission tomography (PET) using 18F-fluorodeoxyglucose (FDG) and computed tomography (CT) will be used. None of the participants were analyzed
Time Frame: FDG PET scan at baseline and Week 2, CT scan at baseline and Week 12
Population: Data were not collected.
Arm/Group | Sunitinib Pill
Number analyzed (Participants) | 0

3. Secondary Outcome: Alteration in Diffusion and Vascularity Kinetics
Description: The Response Evaluation Criteria in Solid Tumors (RECIST) criteria may be insensitive in assessing GIST so the Choi criteria will be used. The Choi criteria accounts for morphologic tumor changes and biologic alterations. Diffusion-weighted magnetic resonance imaging (MRI) and dynamic contrast magnetic resonance will be used to find the vascular permeability and apparent diffusion coefficient 9ACD) at baseline, Week 2 and Week 6. Weeks 2 and 6 values will be compared to the baseline values using paired t tests.
Time Frame: MRI at baseline, Week 2 and Week 6
Population: Data were not collected
Arm/Group | Sunitinib Pill
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: February 2010 to March 2012
Arm/Group | Sunitinib Pill
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Pill (N=5)
neutropenia (Blood and lymphatic system disorders) | 2 (2)
fatigue (General disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 3 (4)
altered taste (Gastrointestinal disorders) | 2 (2)
mucositis (Gastrointestinal disorders) | 2 (2)
hand and foot syndrome (Nervous system disorders) | 2 (2)
hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1)
hyponatremia (Blood and lymphatic system disorders) | 1 (1)
gastrointestinal reflux disease (Gastrointestinal disorders) | 2 (2)
hypertension (Cardiac disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
swelling (Musculoskeletal and connective tissue disorders) | 1 (1) — lower extremity
nausea (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This Pilot trial was terminated early due sluggish accrual; thereby, resulting in much smaller numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No